CLINICAL TRIAL: NCT02799251
Title: Assessment of Postoperative Lymphopenia as Risk Factor for Postoperative Infections: EVALYMPH Study
Brief Title: Assessment of Postoperative Lymphopenia as Risk Factor for Postoperative Infections
Acronym: EVALYMPH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1600010
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cancer of the Digestive System; Thoracic Diseases
Keywords: lymphopenia; postoperative infection; thoracic cancer surgery; digestive cancer surgery
MeSH Terms: conditions — Digestive System Neoplasms; Thoracic Diseases; Lymphopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collection of plasma cell rate: Post operative infections and their association with lymphopenia are assessed in this study for patients over 18 years of age undergoing digestive or thoracic cancer surgery under general anesthesia.
  Interventions: Other: Collection of plasma cell rate

INTERVENTIONS:
Other: Collection of plasma cell rate — Lymphocytes counts are obtained from patients undergoing pulmonary or digestive cancer surgery. The rates are assessed before surgery (day 0) and at days 1, 3, 5 and 8 after surgery. Anesthetic and surgical procedures are collected as well as risk factors for postoperative infections recognized in the literature. Clinical and biological signs of infection are collected.

SUMMARY:
Postoperative infections are one of the most common complications in thoracic and digestive cancer surgery. Former studies have demonstrated that inflammatory response is altered during peri-operative period causing lymphopenia. It has been suggested that lymphopenia may contribute to postoperative infection. To date, no one has proved it in a multivariate analysis. The aim of this study is to determine if lymphopenia is associated with postoperative infections in thoracic and digestive cancer surgery.

DETAILED DESCRIPTION:
Postoperative infections are one of the most common complications in thoracic and digestive cancer surgery. Former studies have demonstrated that inflammatory response is altered during peri-operative period causing lymphopenia. It has been suggested that lymphopenia may contribute to postoperative infection. To date, no one has proved it in a multivariate analysis.

The aim of this study is to determine if lymphopenia is associated with postoperative infections in thoracic and digestive cancer surgery. It is a multicenter French cohort study. Lymphocytes counts are obtained from patients undergoing pulmonary or digestive cancer surgery before surgery (day-0) as well 1, 3, 5 and 8 days after surgery. Anesthetic and surgical procedures are collected as well as risk factors for postoperative infections recognized in the literature. Clinical and biological signs of infection are collected.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing digestive or thoracic cancer surgery under general anesthesia.

Exclusion Criteria:

* pregnant women,
* malignant blood disease,
* allograft patient,
* preoperative sepsis or preoperative systemic inflammatory response syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age undergoing digestive or thoracic cancer surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Presence of post operative infection | 1 month
  Patients undergoing general anesthesia for thoracic or digestive surgery could present lymphopenia. In this situation, the presence of post operative infection is notified. The correlation between lymphopenia and post operative infections is studied.

SECONDARY OUTCOMES:
Anesthetic and surgical parameters | 1 month
  To identify anesthetic and surgical parameters influencing postoperative lymphocytes cells count.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Molliex, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (20):
- France (20):
  - Chu Angers, Angers
  - Hôpital Côtes de Nacre CHU CAEN, Caen
  - Hôpital Estaing CHU CLERMONT-FERRAND, Clermont-Ferrand
  - Hôpital Beaujon CHU PARIS 1, Clichy
  - Hôpital Michallon CHU GRENOBLE, La Tronche
  - Hôpital Huriez CHRU LILLE, Lille
  - Hôpital Edouard Herriot CHU LYON, Lyon
  - Hôpital La croix Rousse CHU LYON, Lyon
  - Hôpital Lyon Sud CHU LYON, Lyon
  - Hôpital Nord CHU MARSEILLE, Marseille
  - Hôpital La Timone CHU MARSEILLE, Marseille
  - Hôpital Hôtel-Dieu CHU NANTES, Nantes
  - Hôpital Carémeau CHU NIMES, Nîmes
  - Hôpital Saint Louis-Lariboisière CHU PARIS 5, Paris
  - Hôpital Saint-Antoine CHU PARIS 4, Paris
  - Hôpital La pitié-Salpetrière CHU PARIS 3, Paris
  - Hôpital Bichat CHU PARIS 2, Paris
  - Hôpital Pontchaillou CHU RENNES, Rennes
  - Hôpital Central CHRU STRASBOURG, Strasbourg
  - Centre de Lutte contre le Cancer, TOULOUSE, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petit L, Pastene B, Dupont G, Baffeleuf B, Goulevant PA, Fellahi JL, Gricourt Y, Lebuffe G, Ouattara A, Fischer MO, Mertes PM, Eyraud D, Bouhemad B, Gomola A, Montravers P, Alingrin J, Flory L, Incagnoli P, Boisson M, Leone M, Monneret G, Lukaszewicz AC, Pereira B, Molliex S; for the EVALYMPH study group. Postoperative lymphopaenia as a risk factor for postoperative infections in cancer surgery: A prospective multicentre cohort study (the EVALYMPH study). Eur J Anaesthesiol. 2025 Mar 1;42(3):244-254. doi: 10.1097/EJA.0000000000002089. Epub 2024 Oct 29. PMID 39474711